CLINICAL TRIAL: NCT03877783
Title: Diet, Physical Exercise and Metabolic Control (DEMAND) Intervention to Reduce the Incidence of Major Neurocognitive Disorders Among Individuals With Type 2 Diabetes Combined With Mild Neurocognitive Impairment - a Pilot Study
Brief Title: DEMAND - Multifactorial Study to Reduce Dementia in People With Type 2 Diabetes
Acronym: DEMAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Olov Rolandsson, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DEMAND pilot
Record Dates: First submitted 2019-02-08; First posted 2019-03-18 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes Mellitus; Mild Cognitive Impairment
Keywords: mediterranean diet; physical fitness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group of intervention (Experimental): participants receive
  1. personalized advice of a dietician about mediterranean diet
  2. individualized training program,
  3. recommendation about optimized pharmacological treatment as in high risk groups for cardiovascular diseases
  Interventions: Dietary Supplement: mediterranean diet; Behavioral: individualized fitness program; Other: recommended modified pharmacological treatment
- group of control (No Intervention): participants receive
  1. written information about the advantages of a healthy diet
  2. written information about the advantages of physical activity,
  3. medical treatment according to the latest version of the national guidelines issued by the Swedish Medical Product Agency

INTERVENTIONS:
Dietary Supplement: mediterranean diet — The recommended Mediterranean diet is based on lean meat, fish, eggs, vegetables, fruits, berries, and nuts. Extra-virgin olive oil is the recommended additional fat source for use in food preparation and dressings. Recommended exclusions or restrictions include dairy products, cereals, added salt, refined fats, and sugar. Participants in the intervention group will receive weekly deliveries of olive oil and mixed nuts, free of cost, and they will receive recipes for Mediterranean meals on a regular basis. During the study, the intervention group will receive written, personalized advice from a project dietician on how to improve their Mediterranean diets. This written personalized advice will be based on the reported food intake, its coherence with a Mediterranean diet, and its adherence to the recommended intakes of energy and nutrients for each participant.
  Arms: group of intervention
Behavioral: individualized fitness program — The exercise intervention will consist of individualized training programs designed to improve cardiovascular fitness (VO2). A personal trainer will distribute the training program instructions and monitor the training during the entire intervention. Support will be provided via text messages. The training intensity will be based on results from an extensive pre-test of individual physical fitness performance, and we will adjust the intensity over the study period, as fitness improves. The goal is to engage participants in training three times per week, for up to one hour per training session. The individualized training programs will consist of brisk walks, jogging, and cycling, tailored to each participant. To ensure that the training intensity is sufficient to improve cardiovascular fitness, heart rate will be monitored during each session.
  Arms: group of intervention
Other: recommended modified pharmacological treatment — Hyperglycemia: first metformin till target level of HbA1c 1) 53-58 mmol/mol for patients with ≤2 coexisting chronic illnesses or 2) 59-64 mmol/mol for those with established cardiovascular disease (CVD). We will recommend a second glucose-lowering drug when HbA1c is not achieved and which reduce CVD even when the participant does not have a manifest CVD.
  Hypertension: will be treated to achieve a target level according to European guidelines. Start with a combination of a renin-angiotensin system (RAS)-blocker and a thiazide in low dose or a combination of a RAS-blocker a calcium channel blocker in low dose. If the target is not reached within 12 weeks additional drugs should be added.
  Dyslipidemia: Patients with a CVD risk of 2-8% within 5 years should receive treatment with atorvastatin 10mg +ezetimib 10mg; CVD risk 8-20%, atorvastatin 20mg + ezetimib 10mg and CVD risk > 20% atorvastatin 40-80mg +ezetimib 10mg.
  Arms: group of intervention

SUMMARY:
In the DEMAND pilot study, we will recruit and randomize 80 participants at two study sites (Umeå and Uppsala) for a one-year intervention. The primary objectives are to study the inclusion rate, the adherence rate, and the acceptability of the intervention. The secondary objectives are to examine the effect of the intervention on intermediate outcomes, including metabolic control (i.e., blood glucose and lipids), body weight, blood pressure, physical fitness, and cognitive function. Third, the investigators will perform focus group interviews to explore the participants views on the intervention to assess the acceptability. The interventions include (a) Mediterranean diet (b) an individualized physical training program and (c) pharmacological treatment for type 2 diabetes (T2D) aimed to achieve individualized optimal goals, according to national guidelines, taking into account the risk of hypoglycaemia. This multi-component intervention is more comprehensive than usual care, and it specifically focuses on vascular domains.

DETAILED DESCRIPTION:
To be inserted.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes diagnosed in the last year
* age >=65 years
* signed consent form
* Mild cognitive impairment

Exclusion Criteria:

* diagnosis type 1 diabetes
* major neurocognitive degeneration
* serious illness with live expectancy less than 3 years
* drug- or alcohol-abuse or other neurological / psychiatric illness which affects the outcome
* depressive syndrome
* predicted inability to conduct the study because of drug abuse, serious illness, language issues
* documented episodes of hypoglycemia where help of a third part was needed
* Allergy to fish or nuts
* Angina pectoris
* Heart failure (NYHA 3-4)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
inclusion rate | 4 months
  How many subjects (n) will be randomized within four months?
adherence rate | 1 year
  What is the proportion (%) of subjects in the intervention group who will adhere to 90% of the diet, exercise and medical intervention?
retention rate | 1 year
  What is the proportion of drop-out in the two groups?

SECONDARY OUTCOMES:
Metabolic change | 1 year
  Is there a significant decrease in HbA1c, blood pressure, and blood lipids in the intervention group compared to the control group?
Memory function | 1 year
  Is the decline in memory function lower in the intervention froup compared to the control group?

CONTACTS AND LOCATIONS:
Overall Officials: Olov Rolandsson, Professor, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Västerbotten County, Sweden